CLINICAL TRIAL: NCT03371368
Title: Metabolic and Endocrine Effects of Bariatric Surgery
Brief Title: Metabolism and Bariatric Surgery Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Judith Korner, Professor of Medicine at the Columbia University Medical Center, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAR3662; R01DK072011 (NIH)
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Insulin Resistance; Obesity
Keywords: Obesity; Insulin Resistance; Bariatric Surgery; Gastric Bypass; Sleeve Gastrectomy
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Intervention Model Description: Cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Gastric Bypass Diabetic and Non-diabetic (Other): Roux-en-Y gastric bypass surgery
  Interventions: Procedure: Roux-en-Y Gastric Bypass (RYGBP)
- Sleeve Gastrectomy Diabetic and Non-diabetic (Other): sleeve gastrectomy surgery
  Interventions: Procedure: Sleeve Gastrectomy (SG)
- Very Low Calorie Diet Diabetic and Non-diabetic (Active Comparator): very low calorie diet
  Interventions: Behavioral: Very Low Calorie Diet (VLCD)
- Obese Control Group (No Intervention): Non-diabetic obese subjects
- Lean Control Group (No Intervention): Non-diabetic lean subjects

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass (RYGBP) — This is a standard RYGBP procedure that would be performed clinically and is not research-specific.
  Other Names: RYGBP
  Arms: Gastric Bypass Diabetic and Non-diabetic
Procedure: Sleeve Gastrectomy (SG) — This is a standard SG procedure that would be performed clinically and is not research-specific.
  Other Names: SG
  Arms: Sleeve Gastrectomy Diabetic and Non-diabetic
Behavioral: Very Low Calorie Diet (VLCD) — Weight loss with calorie restricted liquid diet. Subjects will be placed on a 800 kcal/day diet with a meal replacement (Optifast) provided by the investigator for 12 weeks. Then, transitioning to a higher calorie diet intake up to a year. Subjects will be closely monitored by study dietitian
  Other Names: VLCD
  Arms: Very Low Calorie Diet Diabetic and Non-diabetic

SUMMARY:
The purpose of this study is to determine if diet-induced weight loss causes different changes in hormones that control appetite and glucose control than surgery-induced weight loss. The overall research plan is a non-randomized prospective study of 3 different weight loss (WL) interventions and a lean and an obese healthy control group.

DETAILED DESCRIPTION:
Weight loss (WL) improves obesity-related co-morbidities such as type 2 diabetes mellitus (DM). Unfortunately, WL through life-style interventions has a high degree of relapse and the lack of safe, effective and affordable therapies together with an increase in the prevalence of morbid obesity has led to a rise in bariatric procedures. Clinical trials in patients with DM show that improvements in glycemia vary between procedures and occur in the following order: Roux-en-Y gastric bypass (RYGB) > sleeve gastrectomy (SG) > laparoscopic adjustable gastric banding (LAGB) > medical/life-style therapy. This order mirrors the amount of WL with each intervention and is a major driver of glycemic improvement. The investigators have shown profound changes unique to RYGB and SG in levels of hormones that make up the "gut-brain" and "enteroinsular" axes. The association of some of these hormones with insulin sensitivity (IS) and glycemia, independent of WL strongly suggests that glycemic improvements after surgery occur in part through pathways that are distinct from just calorie restriction. This study builds on results showing that levels of fibroblast growth factor 19 (FGF19), a protein secreted by intestinal cells, are increased after RYGB and SG but not after low calorie diet (LCD). This difference may affect hormones that control the stress response to weight loss. The investigators will explore differences in hormones of the gut that affect appetite, body weight, and stress response in healthy lean and obese individuals. Obese individuals will also be studied before and after 15% body weight loss induced by LCD, RYGB or SG, and again at 1 year after study enrollment.

ELIGIBILITY:
Inclusion Criteria:

Men and women Ages 18-65 Years Old

Exclusion Criteria:

1. Altered Sleep-wake Cycle
2. Type 1 or 2 Diabetes
3. Previous Bariatric Surgery
4. Lactose Intolerance
5. Any Special Diet restrictions.
6. Use of medications that may affect body weight at screening or during a 3-month period prior.
7. Untreated thyroid disease
8. Other medical conditions like Cushing's, acromegaly, Hearth failure, Crohn's disease, etc.
9. Pregnancy
10. Tobacco or opioid use
11. Alcohol dependence
12. > 3% weight change over the 3month period prior to screening
13. Unwillingness to maintain current level of physical activity over duration of study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Change in urine free cortisol level | Baseline and 1 year
  A linear mixed effects model will be used to compare the cortisol changes between the LCD and the surgery groups. Specifically, cortisol change will be modeled as longitudinal outcome, and the main predictors are time and treatment group, and the time-treatment interaction.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Korner, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States